CLINICAL TRIAL: NCT05360771
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study on the Safety and Effectiveness of the SnowyTM PFO Closure System in Plugging Patent Foramen Ovale
Brief Title: Study on the Safety and Effectiveness of the SnowyTM PFO Closure System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Dinova EP Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PFO-001
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Percutaneously occlusion of PFO with SnowyTM PFO closure system
  Interventions: Device: SnowyTM PFO closure system
- control group (Experimental): Percutaneously occlusion of PFO with Cardi-o-fix PFO occluder
  Interventions: Device: Cardi-o-fix PFO occluder

INTERVENTIONS:
Device: SnowyTM PFO closure system — Percutaneously occlusion of PFO with SnowyTM PFO closure system
  Arms: treatment group
Device: Cardi-o-fix PFO occluder — Percutaneously occlusion of PFO with Cardi-o-fix PFO occluder
  Arms: control group

SUMMARY:
To evaluate the safety and effectiveness of the SnowyTM PFO closure system in plugging patent foramen ovale

DETAILED DESCRIPTION:
A prospective, multicenter, randomized controlled clinical trial is conducted to evaluate the safety and effectiveness of PFO closure system produced by Hangzhou Dinova EP Technology Co., Ltd.., Ltd. in closing patent foramen ovale (PFO). 242 patients are expected to be selected. They are randomly divided into the PFO closure system treatment group (121 cases) and the Chinese medicine Shengjie Cardi-o-fix PFO occluder treatment group (121 cases) according to 1:1. All patients will be followed up to 7 days after operation or before discharge, 1 month, 3 month, 6 month, 1 year, 2 year, 3 year, 4 year and 5 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years old, regardless of gender
2. Transthoracic echocardiographic contrast echocardiography (cTTE) confirmed the presence of PFO and at least moderate (see above definition) RLS (in Valsalva active/resting state)
3. Existence of at least one of the following conditions： 1) Unexplained stroke or TIA 2) intractable or chronic migraine
4. The subjects are informed of the nature of the study and agreed to all requirements for participation in the study, signed the informed consent form, and agree to complete the follow-up and follow-up examination

Exclusion Criteria:

1. Patients have definite causes of stroke unrelated to the PFO
2. RLS caused by other causes, such as atrial septal defect or pulmonary arteriovenous shunt
3. Atrial fibrillation or atrial flutter
4. Mitral and aortic stenosis or severe regurgitation
5. Dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy
6. Active endocarditis or other untreated infectious diseases
7. Left ventricular ejection fraction (LVEF) < 40%, or NYHA cardiac function grade III-IV
8. Uncontrollable hypertension
9. Previous intracardiac surgery
10. Myocardial infarction or unstable angina pectoris within 6 months
11. Contraindications to anticoagulants or antiplatelet drugs
12. High risk of bleeding
13. severe liver function impairment（alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of normal value）
14. Serum creatinine greater than 2 times the upper limit of normal or with any history of renal dialysis or renal transplantation
15. Severe pulmonary disease including pulmonary hypertension (clinical diagnosis)
16. Nickel or contrast allergy
17. Active or planned (within 12 months) pregnancy, or lactating female patients
18. Malignant tumors or other serious diseases resulting in a life expectancy of less than 12 months
19. Psychiatric conditions that may interfere with medical compliance and compliance with follow-up
20. Concomitant participation in other clinical trials
21. The investigator determines that the patient is unsuitable because of reasons not listed but thought to interfere with safe trial participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
The success rate of PFO effective occlusion | 6 months after the procedure
  The amount of right to left shunt (RLS) confirmed by imaging examination after occluder implantation is grade 0-I

SECONDARY OUTCOMES:
Number of Participants with Device success | immediately after the procedure
  The successful implantation of occluder is defined as the successful delivery and release of occluder during operation, the position of occluder is appropriate and the morphological structure is normal
Number of Participants with Procedural success | immediately after the procedure
  The occluder is successfully implanted and there are no severe adverse events (SAE) during routine hospitalization. SAE include but are not limited to death, systemic embolism, occluder embolism/displacement, occluder thrombosis, heart injury and perforation, pericardial tamponade / pericardial effusion (pericardial effusion leads to hemodynamic damage or requires pericardiocentesis; prolonged hospitalization for more than 48 hours; hospitalization is required), infective endocarditis, atrial fibrillation, severe vascular access complications
Complete closure rate | 6 months after the procedure
  No RLS is confirmed by imaging examination after occluder implantation
Migraine Headache Impact Test (HIT-6) scores 6 months after operation (compared with baseline) | 6 months after the procedure
  The scores range from 36 to 78 (higher scores mean a worse outcome).
Incidence of serious adverse events | 5 years after the procedure
  Events that cause death or serious deterioration of health conditions during clinical trials, including fatal diseases or injuries, permanent defects in body structure or function, and the need for medical or surgical intervention to avoid permanent defects in body structure or function
Incidence of device-related adverse events | 5 years after the procedure
  Adverse medical events related to the use of devices during clinical trials
All-cause mortality during follow-up | 5 years after the procedure
All-cause stroke during follow-up | 5 years after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China